CLINICAL TRIAL: NCT06656910
Title: The Effect of the Self-compassion Development Program on Bullying and Victimization in Middle School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19/12/23-133; TDK-2024-11388 (Other Grant/Funding Number: Marmara University)
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bullying; Bullying Victimisation
Keywords: bullying; victim; self compassion
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomly assigned intervention and control group, pre-test, post-test after the intervention and follow-up test three months after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervation will be taken.
- Experimental Group (Experimental): In this study, a 7-week self-compassion development program will be implemented on middle school students by a researcher who has a certificate of participation in an 8-week self-compassion development training, a pedagogical formation training certificate, and has experience working as a nurse in a child and adolescent mental health clinic. The content of the program was created by participating in the self-compassion development training and literature review, and expert opinion was obtained.
  Interventions: Behavioral: Self Compassion Group

INTERVENTIONS:
Behavioral: Self Compassion Group — A 7-week self-compassion Programme:
  Course 1:
  Detective Warm-Up Game, Explaining the application of compassion/self-compassion.
  Course 2:
  Draw and Tell Warm-up Game, Breath Awareness Exercise, Mindful Eating Activity.
  Course 3:
  Walking Warm-Up, Body Scan Meditation, How Do You Treat Your Friend Activity.
  Course 4:
  Random Cards warm-up game, Compassion Meditation, Just Like Me Exercise.
  Course 5:
  Break, Self-compassionate letter writing.
  Course 6:
  Tree Drawing Warm-Up Game, Mountain Meditation, Recognize Your Inner Bully, Three Calming Breathing Exercises.
  Course 7:
  Considering the process with participants, Implementation of final tests, Tender farewell.
  Arms: Experimental Group

SUMMARY:
Violence in schools is an important public health problem affecting the health and safety of schools. Peer bullying, which is a common form of school violence, is defined as the behaviour of a bully person or group that deliberately hurts and upsets a person who is weaker than him/her more than once and causes stress in the person exposed to this situation. In peer bullying, there are roles as victim, bully and audience. Bullying has serious consequences on children in all roles. It affects both health and academic success. There are individual, familial, school-related and environmental reasons for peer bullying. There is a significant increase in the rates of peer bullying both in the world and in our country. It is most common in the middle school period among school periods. Self-compassion, a protective factor for individuals, can be expressed as the understanding they show to themselves in the face of negative situations they have encountered throughout their lives. Individuals with self-compassion can approach themselves with love and compassion when they make mistakes or face difficulties in life, thinking that this situation is unique to human beings. When the common characteristics of bullies and victims are examined, it is seen that they experience depression and anxiety, are angry and cannot communicate effectively. Not criticising oneself if it is destructive and cruel, having a compassionate attitude towards oneself protects the individual from negative feelings and thoughts, improves self-esteem and leads to a decrease in depression and anxiety. It is seen that people with high levels of self-compassion exhibit less aggressive behaviour. In this study, a 7-week self-compassion development programme will be implemented for secondary school students.

DETAILED DESCRIPTION:
Peer bullying is a significant school and public health problem that affects school safety and the health of individuals in the school. Peer bullying is a type of aggression in which one or more students intentionally and continuously harass weaker students, and the victim is unable to protect himself. In order for the disturbing situation to be considered peer bullying, there must be an unequal power relationship between individuals, and this situation must be intentional and continuous (Uz, 2018; Olweus, 1999). When the results of recent research and the news in the media are examined, it is seen that violence and bullying incidents in schools, which affect children's academic success and psychological development, are increasing among children and adolescents. According to the 2022 report of the OECD's Programme for International Student Assessment (PISA), on average 20% of students across OECD countries report that they are bullied at least a few times a month. This rate, which was 19% in our country in PISA 2015 data, is reported as 27% according to 2022 data. According to studies, the incidence of peer bullying increases during secondary school (Gökkaya and Sütçü, 2020; Grant et al., 2019; https://pisa.meb.gov.tr/ , Access date: 22/10/2024).

Compassion is to approach failure or error by thinking that it can be a common experience for all people instead of hurting people. Compassion involves being sensitive to other people's sadness, sharing the pain of other individuals, and understanding the people in front of us without judging them. Self-compassion, a protective factor for individuals, can be expressed as the understanding they show themselves in the face of negative situations they encounter throughout their lives. Individuals who show compassion to themselves do not make harsh judgments and self-criticism towards themselves. Self-compassion can also be defined as an individual trying to understand themselves without prejudice, and behaving kindly and compassionately towards themselves instead of judging or criticizing themselves harshly. Self-compassion has three basic components: self-kindness, perception of common human experience, and awareness (Kurtoğlu and Başgül, 2021). Not criticizing oneself if one is destructive and cruel, and being able to have a compassionate attitude towards oneself protects the individual from negative feelings and thoughts, improves self-esteem, and causes a decrease in depression and anxiety (Germer and Neff, 2019). In a study evaluating psychological well-being in the adolescent population, it was observed that there was a significant negative relationship between stress, anxiety, depression levels and self-compassion levels in adolescents (Marsh et al., 2018). There are other studies supporting the fact that individuals with high self-compassion levels exhibit less aggressive attitudes towards other people (Fresnics and Borders, 2017; Sommerfeld and Bitton, 2020). Individuals who cannot show self-compassion have difficulty developing appropriate understanding in the painful experiences of others (Saricaoğlu and Arslan, 2019). When the information obtained from the literature is evaluated, it is thought that the self-compassion development program will have an effect on middle school students' bullying and victimization.

The research was planned as a randomly assigned intervention and control group, pre-test, post-test after the intervention and follow-up test three months after the intervention. The data will be collected with Personal Information Form, Identifying Victims of Peer Bullying Scale, Identifying Peer Bullies Scale and Self-Compassion Scale Short Form.

It was aimed to reach a total of 102 students, 51 in the experimental group and 51 in the control group, out of the students enrolled in the 5th grade (N=185) in the Milli Eğitim Vakfı Middle School in Usküdar district of Istanbul province. The participants were assigned to groups by lot.

This study aims to evaluate the effects of a self-compassion development program on bullying and victimization among secondary school students.

ELIGIBILITY:
Inclusion Criteria:

* Being a 5th grade middle school student
* Volunteering to participate in the research
* No vision, hearing, comprehension problems
* Regular attendance to the sessions

Exclusion Criteria:

* Lack of parental permission to participate in the study
* Failure to fill in the forms related to the research completely
* Abandoning the research at any time during the research

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Mean of Peer Bullying and Victimization Score | Baseline (Before the intervention) and from enrollment to the end of intervention 7 weeks and 12 weeks.
  Mean of victimization score will be determined by Identifying Victims of Peer Bullying Scale. The scale, developed by Mynard and Joseph (2000) and adapted to Turkish by Gültekin and Sayıl (2005) for students aged 11-16, consists of 5 sub-dimensions and 27 items. The lowest score that can be obtained from the scale is 0, and the highest score is 54. A high score obtained from the scale indicates that the person is frequently the target of peer attack, while a low score indicates that the person is rarely or never a target.
  Mean of peer bullying score will be determined by Identifying Peer Bullies Scale. This scale developed by Mynard and Joseph (2000) and adapted into Turkish by Gültekin and Sayıl by adding the question "So, how much do you do this behavior?" developed by Pekel and Uçanok (2005). The lowest score that can be obtained from the scale is 0, and the highest score is 54. As the scores obtained from the scale increase, the rate of bully behaviour increases.

SECONDARY OUTCOMES:
Mean of Self Compassion score | Baseline (Before the intervention) and from enrollment to the end of intervention 7 weeks and 12 weeks.
  Mean of Self Compassion score will be determinated Self-compassion scale short form. The Self-Compassion Scale short form was developed by Neff (2003) and adapted into Turkish by Yıldırım and Sarı (2018) to examine the psychometric properties of the scale on adolescents. The scale is a 5-point Likert type, consisting of 11 items and a single dimension. The reliability Cronbach alpha internal consistency coefficient of the scale is 0.75. The 1st, 4th, 8th, 9th, 10th and 11th items on the scale are reverse coded. The highest score that can be obtained from the scale is 55, and the lowest score is 11. A high score obtained from the scale indicates that the individual has a high level of self-compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Milli Eğitim Vakfı Middle School, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yıldırım M, Sarı T. Öz-Şefkat Ölçeği Kısa Formu'nun Türkçe Uyarlaması: Geçerlik Ve Güvenirlik Çalışması. Abant İzzet Baysal Üniversitesi Eğitim Fakültesi Dergisi. 2018; 18(4): 2502-17
- [Result] Pekel NU, Uçanok Z. Akran zorbalığı gruplarında yalnızlık ve akademik başarı ile sosyometrik statüye göre zorba/ kurban davranış türleri. Türk Psikoloji Dergisi.2005; 56: 77-92
- [Result] Mynard H, Joseph S. Development of the multidimensional peer-victimization scale. Aggressive Behavior: Official Journal of the International Society for Research on Aggression.2000; 26(2):169-78
- [Result] Gültekin Z, Sayıl M. Akran Zorbalığını Belirleme Ölçeği geliştirme çalışması. Türk Psikoloji Yazıları. 2005; 15: 47- 61.
- [Result] Uz R. Okullarda Şiddet. 1. Basım, Sentez Yayıncılık. Bursa; 2018
- [Result] Sommerfeld E, Shechory Bitton M. Rejection Sensitivity, Self-Compassion, and Aggressive Behavior: The Role of Borderline Features as a Mediator. Front Psychol. 2020 Jan 24;11:44. doi: 10.3389/fpsyg.2020.00044. eCollection 2020. PMID 32038443
- [Result] Sarıcaoğlu H, Arslan C. Bilinçli öz-anlayış programının üniversite öğrencilerinin öz-anlayışına etkisi. Manas Sosyal Araştırmalar Dergisi. 2019; 8(3), 2381-99
- [Result] Olweus D. In P. K. Smith, Y. Morita, J. Junger-Tas, D. Olweus, R. Catalano & P. Slee (Eds.), The nature of school bullying: A cross national perspective . London and New York: Routledge. 1999 ; 7-27
- [Result] Marsh IC, Chan SWY, MacBeth A. Self-compassion and Psychological Distress in Adolescents-a Meta-analysis. Mindfulness (N Y). 2018;9(4):1011-1027. doi: 10.1007/s12671-017-0850-7. Epub 2017 Nov 25. PMID 30100930
- [Result] Kurtoğlu M, Başgül ŞS. Koruyucu faktör olarak öz-şefkat üzerine bir derleme çalışması. Journal of CognitiveBehavioral Psychotherapy and Research. 2013;10(1): 56-65
- [Result] Grant NJ, Merrin GJ, King MT, Espelage DL. Ortaokul öğrencileri arasında zorbalığa ilişkin aile içi şiddet ve akran sapkınlığının kişi içi ve kişiler arası ilişkilerinin incelenmesi. Şiddet Psikolojisi.2019; 9 (1): 18-27
- [Result] Gökkaya F, Sütçü ST. Akran zorbalığının ortaokul öğrencileri arasında yaygınlığının incelenmesi. Hacettepe Üniversitesi Eğitim Fakültesi Dergisi. 2020; 35(1); 40-54
- [Result] Germer CK, Neff K. Öz Şefkatli Farkındalık Uygulama Rehberi. Çeviren: Tarımtay Altun F. 1. Basım, Diyojen Yayıncılık Ltd. Şti., İstanbul; 2020
- [Result] Fresnics A, Borders A. Angry rumination mediates the unique associations between self-compassion and anger and aggression. Mindfulness.2017; 8(3): 554-64